CLINICAL TRIAL: NCT04617821
Title: A Phase Ⅲ, Randomized Controlled Study to Evaluate the Efficacy and Safety of the Combination of Nab-paclitaxel and Gemcitabine Versus mFOLFIRINOX in Treating Patients With Borderline Reseactable and Locally Advanced Pancreatic Cancer
Brief Title: AG vs mFOLFIRINOX as Neoadjuvant Therapy for Borderline Reseactable and Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Vice President of Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-28
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Borderline Resectable Pancreatic Cancer; Locally Advanced Pancreatic Adenocarcinoma
Keywords: neoadjuvant chemotherapy; albumin bound paclitaxel; mFOLFIRINOX
MeSH Terms: interventions — Taxes; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Three hundred patients with borderline resectable and locally advanced pancreatic cancer are randomized 1:1 to the AG and mFOLFIRINOX chemotherapy groups and to observe the total survival.
Masking Description: open-label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- albumin bound paclitaxel plus gemcitabine (Experimental): Albumin-bound paclitaxel and gemcitabine were given intravenous infusion, repeated every 4 weeks for 1, 8, and 15 days, for a total of 4 to 6 cycles.
  Interventions: Drug: Nab paclitaxel plus gemcitabine
- mFOFLIRINOX (Active Comparator): Intravenous oxaliplatin for 2 hours, day 1;Intravenous infusion of calcium formyl tetrahydrofolate (LV) for 2 h, day 1;Irinotecan intravenous infusion is added 30 minutes later for 90 minutes, day 1;Intravenous infusion of 5-fluorouracil (5-FU) continued for 46 hours.Repeat every 2 weeks for a total of 4-6 cycles.
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Nab paclitaxel plus gemcitabine — Albumin-bound paclitaxel and gemcitabine are given intravenous infusion, repeated every 4 weeks for 1, 8, and 15 days, for a total of 4 to 6 cycle.
  Other Names: AG regimen
  Arms: albumin bound paclitaxel plus gemcitabine
Drug: mFOLFIRINOX — Intravenous oxaliplatin for 2 hours, day 1;Intravenous infusion of calcium formyl tetrahydrofolate (LV) for 2 h, day 1;Irinotecan intravenous infusion is added 30 minutes later for 90 minutes, day 1;Intravenous infusion of 5-fluorouracil (5-FU) continued for 46 hours.Repeat every 2 weeks for a total of 4-6 cycles.
  Other Names: modified FOLFIRINOX regimen
  Arms: mFOFLIRINOX

SUMMARY:
This is a prospective, single-center, randomized, controlled phase Ⅲ study.

DETAILED DESCRIPTION:
Three hundred patients with borderline resectable and locally advanced pancreatic cancer will be randomized 1:1 (150 :150) to the AG and mFOLFIRINOX chemotherapy groups and to observe the overall survival.

The AG regimen: albumin-bound paclitaxel and gemcitabine are given intravenous infusion, repeated every 4 weeks for 1, 8, and 15 days, for a total of 4 to 6 cycles.

MFOLFIRINOX: Intravenous oxaliplatin for 2 hours, day 1;Intravenous infusion of calcium formyl tetrahydrofolate (LV) for 2 h, day 1;Irinotecan intravenous infusion is added 30 minutes later for 90 minutes, day 1;Intravenous infusion of 5-fluorouracil (5-FU) continued for 46 hours.Repeat every 2 weeks for a total of 4-6 cycles.

After neoadjuvant chemotherapy, the surgery will be evaluated according to the patient's tumor and systemic condition.

The first cycle of adjuvant chemotherapy begins 4-8 weeks after radical resection, and the choice of adjuvant chemotherapy regimen depends on the response to neoadjuvant chemotherapy.If neoadjuvant chemotherapy is effective, adjuvant chemotherapy maintains the original regimen.Adjuvant chemotherapy has 4 cycles of treatment.

Relevant examinations were performed before and after each cycle of medication to assess safety events, imaging review was performed every 2 cycles during the treatment period and every 3 months during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥18 years and ≤ 80 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Radiographically confirmed after borderline resectable or locally advanced pancreatic adenocarcinoma.
* No any other anti-tumor therapy prior to neoadjuvant chemotherapy, including intervention chemoembolization, ablation, radiotherapy, chemotherapy and molecular targeted therapy.
* No any other anti-tumor therapy prior to neoadjuvant chemotherapy, including intervention chemoembolization, ablation, radiotherapy, chemotherapy and molecular targeted therapy.
* No serious blood system, heart, lung function abnormalities and immune defects (refer to the respective standards)
* White blood cell (WBC) ≥ 3 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelets (PLT) ≥ 100 × 109/L; Hemoglobin (Hgb)≥ 9 g/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 × institutional upper limit of normal (ULN); Total bilirubin (TBIL) ≤ ULN; Creatinine (CRE) ≤ 1.5 × ULN
* Prothrombin time (PT) and international normalized ratio (INR) ≤ 1.5 ×ULN
* Comply with research visit plans and other program requirements.

Exclusion Criteria:

* with other systemic malignancies
* Patients who were treated with any other anti-tumor therapy prior to neoadjuvant chemotherapy, including intervention chemoembolization, ablation, radiotherapy, chemotherapy and molecular targeted therapy.
* used any other study drug within 7 days prior to enrollment;
* Patients with central nervous system diseases, mental illness, unstable angina pectoris, congestive heart failure, severe arrhythmia and other serious diseases that cannot be controlled
* History of allergic reactions attributed to compounds of similar chemical or biological composition to study drug and alike.
* Patients who are using and expected to use warfarin in long term
* Patients may leave the observation for 14 days or more during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
overall survival | from randomization to death, up to 36 months
  To evaluate the overall survival of patients with borderline resectable and locally advanced pancreatic cancer after treated neoadjuvant chemotherapy

SECONDARY OUTCOMES:
recurrence free survival | from randomization to recurrence, up to 36 months
  To evaluate the recurrence free survival of patients with borderline resectable and locally advanced pancreatic cancer after treated neoadjuvant chemotherapy
objective response rate | up to 36 months
  To evaluate the objective response rate of patients with borderline resectable and locally advanced pancreatic cancer after treated neoadjuvant chemotherapy
resection rate | up to 36 months
  The proportion of patients who become operable from inoperable after neoadjuvant chemotherapy.
R0 resection | up to 36 months
  The proportion of R0 resection among patients who undergo operations.
postoperative complications | up to 36 months
  The incidence of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China